CLINICAL TRIAL: NCT02890043
Title: Clinical Trial for the Application of Tirobot System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: Beijing Tinavi Medical Technology Co Ltd (Unknown); Chinese PLA General Hospital (Other); Tianjin Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, Director, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JST-Tirobot-2016
Record Dates: First submitted 2016-08-21; First posted 2016-09-07 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Fusion of Spine (Disease); Robotic Surgical Procedures
Keywords: spine; robot-assisted surgery; pedicle screw
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot (Experimental): Intervention: Surgery: robot-assisted spine surgery, device: TiRobot surgery system
  Interventions: Procedure: robot-assisted spine surgery; Device: TiRobot system
- Free-hand (Active Comparator): Intervention: Surgery: free-hand surgery
  Interventions: Procedure: free-hand surgery

INTERVENTIONS:
Procedure: robot-assisted spine surgery — robot-assisted spine surgery using Tirobot system
  Arms: Robot
Procedure: free-hand surgery — traditional free-hand surgery
  Arms: Free-hand
Device: TiRobot system — a robot-assisted spine surgery system
  Arms: Robot

SUMMARY:
The object of this study was to evaluate the accuracy and safety of the Tirobot system.

DETAILED DESCRIPTION:
Tirobot system is a new-type medical robot-assisted surgery system that designed for spine and traumatic orthopaedic surgeries. This system has been certified by CE. The accuracy and safety of pedicle screw placement using this system will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* traumatic or degenerative thoracolumbar disease required for pedicle screw fixation surgery

Exclusion Criteria:

* severe osteoporosis
* old thoracolumbar fracture
* deformity of pedicle
* combined with coagulation disorders
* combined with other systematic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
perforation rate of pedicle screws | up to postoperative 3 days
  number of pedicle screws breaching out pedicles on postoperative CT image/ total screw number

SECONDARY OUTCOMES:
operation time | through the operation complete, an average of 2 hours
  total operation time of the surgery (time in minutes)
complications | up to postoperative 3 months
  Number of Adverse Events That Are Related to Treatments

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, MD, Study Chair — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498
- [Result] Karapinar L, Erel N, Ozturk H, Altay T, Kaya A. Pedicle screw placement with a free hand technique in thoracolumbar spine: is it safe? J Spinal Disord Tech. 2008 Feb;21(1):63-7. doi: 10.1097/BSD.0b013e3181453dc6. PMID 18418139
- [Result] Weinstein JN, Rydevik BL, Rauschning W. Anatomic and technical considerations of pedicle screw fixation. Clin Orthop Relat Res. 1992 Nov;(284):34-46. PMID 1395312
- [Derived] Han X, Tian W, Liu Y, Liu B, He D, Sun Y, Han X, Fan M, Zhao J, Xu Y, Zhang Q. Safety and accuracy of robot-assisted versus fluoroscopy-assisted pedicle screw insertion in thoracolumbar spinal surgery: a prospective randomized controlled trial. J Neurosurg Spine. 2019 Feb 8;30(5):615-622. doi: 10.3171/2018.10.SPINE18487. Print 2019 May 1. PMID 30738398